CLINICAL TRIAL: NCT07360509
Title: Evaluation of Treatment Outcomes With Palatal Plate Versus Conventional Tooth Borne Anchorage in Class III Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Yousra Mohamed Saad, principal investigator, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO-109-3-G
Record Dates: First submitted 2026-01-10; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Skeletal Class III Malocclusion
MeSH Terms: interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment of skeletal class III by maxillary advancement using transpalatal arch (Experimental): treatment of skeletal class III by maxillary advancement, using transpalatal arch and facemask
  Interventions: Device: treatment of skeletal class III by maxillary advancement using transpalatal arch and face mask
- treatment of skeletal class III by maxillary advancement by skeletal anchorage (Experimental): treatment of skeletal class III by maxillary advancement by skeletal anchorage using palatal plate and face mask
  Interventions: Device: treatment of skeletal class III by maxillary advancement using palatal plate and face mask

INTERVENTIONS:
Device: treatment of skeletal class III by maxillary advancement using transpalatal arch and face mask — TPA group
  Arms: treatment of skeletal class III by maxillary advancement using transpalatal arch
Device: treatment of skeletal class III by maxillary advancement using palatal plate and face mask — palatal plate group
  Arms: treatment of skeletal class III by maxillary advancement by skeletal anchorage

SUMMARY:
evaluation of treatment outcomes with palatal plate versus conventional tooth borne anchorage in class III patients

DETAILED DESCRIPTION:
group (A) patients were treated with transpalatal arch and facemask. group(B) patients were treated by palatal plate and facemask

ELIGIBILITY:
Inclusion Criteria:

* skeletal class III malocclusion deficient maxilla+ growing patient

Exclusion Criteria:

* adult patient, cleft patient

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
skeletal and dental maxillary changes including SN angle, SNB angle, ANB angle | 3-12 months
  lateral cephalometry

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry , Al Azhar University, Girls Branch, Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Treatment effects of maxillary protraction with palatal plates vs conventional tooth-borne anchorage in growing patients with Class III malocclusion — https://pubmed.ncbi.nlm.nih.gov/35933257/